CLINICAL TRIAL: NCT01719185
Title: A Pilot Study to Assess Whether the Combination of Phentermine and B12 Has a Significant Effect on Weight Loss Among an Obese Study Population
Brief Title: The Effect of Phentermine and B12 on Weight Loss Among Obese Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dr. Michael Lang (Other)
Responsible Party: Sponsor-Investigator, Dr. Michael Lang, Michael Lang, MD, Internal Medicine, Psychiatrics, East Carolina University
Organization: East Carolina University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-001323
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Phentermine; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phentermine and B12 (Experimental): Those in the experimental group will take 37.5 mg of phentermine daily as well as receive 1000 mg intramuscular injections of B12 weekly.
  Interventions: Drug: Phentermine and B12
- Phentermine (Active Comparator): Those in the control group will take phentermine 37.5 mg daily as well as receive 1000 mg intramuscular injections of saline weekly.
  Interventions: Drug: Phentermine

INTERVENTIONS:
Drug: Phentermine and B12
  Other Names: Adipex-P, Cyanocobalamin
  Arms: Phentermine and B12
Drug: Phentermine
  Other Names: Adipex- P
  Arms: Phentermine

SUMMARY:
This is a pilot study designed to test the hypothesis that the combination of phentermine and B12 will result in significantly greater weight loss among obese patients compared to phentermine alone.

DETAILED DESCRIPTION:
This pilot study is a double blind, randomized controlled trial designed to determine the significance of the combination therapy of phentermine and B12 injections among the obese population. The study population will be recruited from the ECU Physicians Internal Medicine clinic. Physicians will select patients meeting inclusion and exclusion criteria from their clinic to be approached for recruitment. Approximately 30 patients will be recruited and blindly randomized to either the treatment group (phentermine and B12 in combination) or the control group (phentermine alone). Patients will be randomized by means of block randomization in a 1:1 ratio. Neither patients nor study team members will be aware of group assignments through the entire duration of the study. Once randomized, both groups will begin taking 37.5 mg/day orally of phentermine as well as receive weekly intramuscular injections of either 1000 mg B12 or Saline depending on their group assignment. The study will consist of approximately 15 visits over the course of 3 months.

ELIGIBILITY:
Individuals can participate in the study if they meet the following inclusion criteria:

* Are over the age of 18
* Have a BMI between 30 and 40
* Have a controlled blood pressure
* Do not have a B12 deficiency
* Are willing to take birth control (if female and not sterile or through menopause)
* Are English speaking

Individuals should not participate in if any of the following apply to them:

* Are not over the age of 18
* Do not have a BMI between 30 and 40
* Do not have a controlled blood pressure
* Have a B12 deficiency
* Females who are pregnant, trying to get pregnant, or not willing to use a method of birth control to ensure they do not become pregnant
* Individuals who do not speak English
* Individuals currently taking Adderall, Ritalin, or any other stimulant medication
* Individuals who have taken phentermine more than once in the past, or within 3 months of study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Weight Change | 24 weeks (6 months)
  Weight change from baseline to 6 weeks, 12 weeks, and 24 weeks among the intervention (phentermine and B12) and control (phentermine) groups.

SECONDARY OUTCOMES:
Blood Pressure | 24 weeks
  Blood pressure changes from baseline to 6 weeks, 12 weeks, and 24 weeks among the intervention and control groups.
Waist Circumference | 24 weeks
  Changes in waist circumference from baseline to 12 weeks and 24 weeks among the intervention and control groups.
Waist to hip ratio | 24 weeks
  Changes in waist to hip ratio from baseline to 12 weeks and 24 weeks among the intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Lang, MD, Principal Investigator — ECU Physicians General Internal Medicine, Psychiatry; James Powell, MD, Study Chair — ECU Physicians General Internal Medicine
Locations (1):
- Brody Outpatient of Brody Medical Sciences Module D, Greenville, North Carolina, United States